CLINICAL TRIAL: NCT06619886
Title: Early Clinical Study to Evaluate the Safety and Efficacy of TP53 R248Q Mutation-specific TCR-T Cell Therapy for Advanced Solid Tumor
Brief Title: TP53 R248Q TCR-T Cell Therapy for Advanced Solid Tumor
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qi Li, Shanghai General Hospital, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP53-R248Q-PC
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumor, Adult; Lung Adenocarcinoma; Pancreas Cancer; Colorectal Cancer; Other Solid Tumor
Keywords: TP53-R248Q; TCR-T; advanced solid tumor
MeSH Terms: conditions — Adenocarcinoma of Lung; Pancreatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TP53 R248Q specific TCR transduction T cell therapy (Experimental): Dose Escalation of TCR T cell product
  Interventions: Biological: Autologous, engineered T Cells targeting TP53 R248Q

INTERVENTIONS:
Biological: Autologous, engineered T Cells targeting TP53 R248Q — TP53-R248Q mutant TCR-T Cells Injection, 28 days as a treatment cycle (cycle number N≤3), each cycle was divided into three D0, D7, D14 infusion, a total of 3 dose groups were set up, the single infusion of cells within the range of ±20% all meet the requirements

SUMMARY:
To evaluate the safety and efficacy of T cell therapy with mutated TP53 R248Q specific TCR transduction in patients with advanced solid tumor expressing the TP53 R248Q mutation and the HLA-A*11:01 allele.

DETAILED DESCRIPTION:
Malignant tumors are a major disease threatening the health of the Chinese people, with about 4.6 million new cancer patients and 2 million deaths each year in China. P53 gene mutation is an important driver gene in the pathogenesis of malignant tumors. P53 gene mutation is present in about half of cancer patients. Tumors carrying P53 gene mutation are insensitive to treatment, have poor response, are easy to be resistant, are easy to relapse, and have a high mortality rate. At present, there is no drug that directly targets P53 gene mutation. Our laboratory has previously built a TCR-T cell R & D platform. Using this platform, we have successfully developed a TCR-T cell specific killing function for tumor cells targeting the R248Q mutation of the most common TP53 protein in hematological tumors and targeting the most high-frequency HLA-A11:01 subtype of TCR-T cells in the Chinese population using in vitro and in vivo animal models, and applied for a Chinese invention patent and PCT invention patent. The findings provide new ideas and treatment methods for immune cell therapy of malignant tumors. At present, we cooperate with the hematology clinical team of Shanghai First People's Hospital and Shanghai Pharmaceutical Group Biotherapy Technology Co., Ltd. to prepare to carry out investigator-initiated clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. signed a written informed consent form (ICF), and can comply with protocol-specified visits and related procedures;
2. aged ≥ 18 years, and ≤ 75 years, male or female;
3. Subject must be pathologically confirmed with one of the histology below:

   Lung carcinoma Colorectal adenocarcinoma Pancreatic adenocarcinoma Any other solid tumor (progression after receiving standard treatment);
4. subjects with TP53R248Q mutation in genetic testing, as determined by DNA or RNA sequencing methods;
5. if patients with brain metastases are asymptomatic and less than 3 brain lesions less than 3 cm in diameter, they may be eligible;
6. ECOG score 0-1;
7. Expected survival of no less than 12 weeks;
8. According to RECISTv1.1 and mRECIST, subjects have at least 1 measurable lesion (lesions that have received local therapy such as radiotherapy and interventional therapy cannot be used as measurable lesions unless imaging evidence confirms that the lesion has clearly progressed), RECISTv1.1 is non-lymph node lesions with the longest diameter ≥ 10 mm on CT or MRI, and/or lymph node lesions with the short diameter ≥ 15 mm; mRECIST is non-lymph node measurable lesion criteria that meet RECISTv1.1 criteria, and showed intratumoral arterial enhancement in enhanced CT or MRI;
9. subjects should provide fresh tumor tissue samples that meet the requirements or within 2 years before signing the ICF;
10. Adequate organ and bone marrow function as defined by the following laboratory criteria: (1) bone marrow function: absolute neutrophil count (ANC) ≥ 1.5 × 109/L; platelet (PLT) ≥ 75 × 109/L (transfusion or hematopoietic stimulating factor not acceptable within 14 days prior to Screening); (2) hemoglobin ≥ 90 g/L; (3) liver function: total bilirubin ≤ 2.5 × ULN; alanine aminotransferase ≤ 5 × ULN; aspartate aminotransferase ≤ 5 × ULN; (4) renal function: serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 60 mL/min (calculated using the Cockcroft-Gault formula); (5) coagulation function: international normalized ratio (INR) ≤ 1.5 × ULN, activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (INR between 2.0 and 3.0 is required for subjects receiving prophylactic anticoagulant therapy);
11. Males of childbearing potential and females of childbearing potential must agree to use effective contraception from signing the ICF until one year after the last cell infusion and females of childbearing potential must have a negative blood pregnancy test at screening.

Exclusion Criteria:

1. previous bone marrow or organ transplantation (including but not limited to liver transplantation) or waiting for transplantation;
2. previous or concurrent history of other malignancies (cured and at least 2 years before screening without recurrence of cervical carcinoma in situ, non-invasive basal cell or squamous cell skin cancer or radical treatment of local prostate cancer, radical resection of ductal carcinoma in situ can be enrolled in the study);
3. hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and HBV DNA > 500 IU/mL (lower limit of detection < HBV DNA ≤ 500 IU/mL, clear lymphocyte conditioning medication before the need for at least 14 days of antiviral therapy and continuous antiviral therapy during the study can be enrolled); hepatitis C virus (HCV) antibody positive and HCV RNA positive; human immunodeficiency virus (HIV) antibody positive; syphilis antibody positive;
4. HLA antibody positive subjects, including weak positive, positive and strong positive (those with different HLA typing sites from TP53R248QTCR-T cell injection can be enrolled in the study);
5. previous treatment with other cell products or TP53 targeted drugs;
6. treatment with any fluorouracil chemotherapeutic drugs or small molecule targeted drugs within 14 days or 5 half-lives (whichever is shorter) before screening, and any antineoplastic biological agents or non-fluorouracil chemotherapeutic agents; radical radiotherapy or extensive radiotherapy within 28 days before screening (except palliative radiotherapy for non-target lesions performed locally to relieve symptoms); traditional Chinese medicine/Chinese herbal medicine and local interventional therapy with antineoplastic indications within 14 days before screening;
7. adverse events caused by previous antineoplastic therapy have not yet recovered to grade 1 or baseline levels, except for alopecia, grade 2 peripheral neurotoxicity, and hypothyroidism stabilized by hormone replacement therapy;
8. live attenuated vaccination within 28 days before screening, or live attenuated vaccination during the study;
9. major surgical treatment (except liver mass biopsy) within 28 days before screening, or major surgical treatment during the study;
10. Requirement for chronic systemic corticosteroids (at doses ≥ 10 mg/day prednisone or equivalent) or other immunosuppressive medication within 14 days prior to the first study drug infusion or during the study, with the exception of inhaled or topical use;
11. Subjects with fungal, bacterial, viral, tuberculosis or other infection requiring systemic anti-infective therapy within 14 days prior to screening;
12. Patients with active or previous autoimmune diseases that may relapse, such as systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vasculitis, psoriasis, etc.;
13. Previous or current interstitial lung disease, dust disease, radiation pneumonitis, severely impaired pulmonary function and other conditions;
14. Third space effusion that is not clinically well controlled before screening, such as pleural effusion and ascites that cannot be controlled by drainage or other methods;
15. History of serious cardiovascular and cerebrovascular diseases, including but not limited to:

    * severe heart rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, grade II-III atrioventricular block, etc.;
    * prolonged QT interval corrected by Fridericia formula (QTcF), > 450 ms in men and > 470 ms in women;
    * acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other ≥ Grade 3 cardiovascular and cerebrovascular events within 6 months before screening;
    * presence of heart failure with New York Heart Association (NYHA) functional class ≥ II or left ventricular ejection fraction (LVEF) < 50%;
    * clinically uncontrolled hypertension, systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg.
16. Patients with a history of pulmonary embolism or severe lower extremity deep venous thrombosis, need to undergo inferior vena cava filter placement and other interventional therapy or need to use therapeutic doses of anticoagulants during screening;
17. Subjects are participating in other interventional clinical studies;
18. Pregnant or lactating women;
19. Researchers believe that subjects have other conditions that may affect compliance or are not suitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-09-24 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Short term Safety of TP53-R248Q TCR-T cell injection in subjects with unresectable, advanced, and/or metastatic solid tumors | 28 days after infusion
  Incidence of dose-limiting toxicities (DLTs) after the infusion of TP53-R248Q TCR-T cell injection;
Long term Safety of TP53-R248Q TCR-T cell injection in subjects with unresectable, advanced, and/or metastatic solid tumors | 28 days after infusion and up to 24 months after infusion
  Incidence of adverse events and serious adverse events; Treatment-emergent adverse events, and serious adverse events

SECONDARY OUTCOMES:
Preliminary anti-tumor activity of TP53-R248Q TCR-T cell injection in subjects with unresectable, advanced, and/or metastatic solid tumors | Up to 24 months after infusion
  Objective Response Rate (ORR) per RECIST V1.1 determined by Investigator assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Qi Li, Prof., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Department of Oncology, Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No